CLINICAL TRIAL: NCT03511248
Title: Investigation of Dietary Nitrate Optimisation by Hyperuricaemia Stratification in Heart Failure
Brief Title: Effect of Dietary Nitrate Ingestion in Heart Failure
Acronym: DiNOmo-HF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: abandoned
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17/LO/1624
Record Dates: First submitted 2018-03-29; First posted 2018-04-27 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Heart Failure, Systolic
Keywords: Heart Failure; Heart Failure with Reduced Ejection Fraction; Nitric Oxide; Inorganic Nitrate
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic

STUDY DESIGN:
Intervention Model Description: Randomised double-blind placebo-controlled parallel two-limb study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind study, with randomisation undertaken by Barts Cardiovascular Clinical Trials Unit
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate-rich Beetroot Juice (Experimental): Individuals will receive a once daily dose of dietary nitrate in the form of a beetroot juice concentrate (70mL) containing ~5-6mmol inorganic nitrate (James White Drinks, UK) for 12 +/- 2 weeks. This dose has been chosen due to several reports demonstrating efficacy in patients with cardiovascular disease.
  Interventions: Dietary Supplement: Nitrate-rich Beetroot Juice
- Nitrate-deplete Beetroot Juice (Placebo Comparator): The placebo control is an identical juice from which the nitrate anion has been removed using a standard anion exchange resin. Visually there is no detectable difference between the juices and previous spectral, ion concentration, sugar levels, ascorbate analysis and taste testing has confirmed no differences in colour and constituents. The process to extract nitrate from the juice is the same technique used to remove inorganic nitrate from general drinking water supplies, and has been approved for use by Ethics Committees. The nitrate-free juice is not considered a drug or medicine, and is classified as a foodstuff.
  Interventions: Dietary Supplement: Nitrate-deplete Beetroot Juice

INTERVENTIONS:
Dietary Supplement: Nitrate-rich Beetroot Juice — The beetroot juice contains approximately 100kcal per 100mL of juice, equivalent to a glass of orange juice; the volume of juice per day for the study is 70mL. Volunteers will be informed that an average woman weighing 65kg should not consume more than 2000kcal per day, and an average man of 75kg not more than 2500kcal per day.
  Arms: Nitrate-rich Beetroot Juice
Dietary Supplement: Nitrate-deplete Beetroot Juice — The beetroot juice contains approximately 100kcal per 100mL of juice, equivalent to a glass of orange juice; the volume of juice per day for the study is 70mL. Volunteers will be informed that an average woman weighing 65kg should not consume more than 2000kcal per day, and an average man of 75kg not more than 2500kcal per day.
  Other Names: Placebo
  Arms: Nitrate-deplete Beetroot Juice

SUMMARY:
This study evaluates the addition of inorganic dietary nitrate to the optimal treatment of patients diagnosed with heart failure with reduced ejection fraction. Some vegetables contain large amounts of inorganic nitrate, and research suggests that this nitrate has beneficial effects on the heart and blood vessels. We have shown in lab experiments that nitrate has positive effects on the heart. We wish to test whether dietary nitrate might be useful in halting deterioration and/or improving heart function in patients with heart failure, with a specific focus on a marker of poor outcome in heart failure: high uric acid levels. Half of the patients will receive nitrate-rich beetroot juice, and the other half a nitrate-deplete placebo beetroot juice.

DETAILED DESCRIPTION:
Background: Heart failure (HF) affects 1-2% of those under 70 years, and 10-20% of those over 70 years in developed countries; approximately 900,000 people in the UK suffer with HF. Despite several promising pre-clinical targets, clinical translation has been disappointing, with very few successful phase 3 studies of new HF therapeutics. Dysfunction of the classical pathways that underlie endothelial nitric oxide (NO) production, with deficient cardiac constitutive NO supply, are thought to play a major role in the pathogenesis of HF. It has been mooted that novel strategies that replace/restore this diminished NO have therapeutic potential.

The organic nitrates, as a method of NO delivery, provide an efficacious treatment in the acute HF setting. However, the development of tolerance, tachyphylaxis, and endothelial dysfunction with long-term use severely limits their utility in chronic heart disease. Alternative methods for sustained NO delivery without tolerance are therefore of interest.

Recent clinical research demonstrates that inorganic nitrate offers this possibility through sequential chemical reduction, first via the enterosalivary circuit to nitrite, and subsequently from nitrite to NO. In particular, pre-clinical research suggests that delivery of NO via this pathway imparts benefit in HF models. Dietary inorganic nitrate is known to provide a safe and non-invasive method to elevate NO in humans, and a once daily dose (5-6mmol), in the form of a beetroot juice, can improve vascular function and reduce blood pressure in hypertensives.

Inorganic nitrate as a HF treatment is particularly exciting since a key pathway involved in the generation of NO from nitrate is xanthine oxidoreductase (XOR); an enzyme upregulated in HF. Conventionally, XOR is considered detrimental as it generates superoxide and uric acid; both exert negative effects on cardiac function, and are associated with worse outcomes in HF. However, XOR also plays an important role in the second step of nitrate bioactivation: conversion of nitrite to NO in the heart. Importantly, we have hypothesised that in an environment of elevated XOR activity, such as HF, delivery of inorganic nitrate to the body would result in reductions in superoxide/uric acid with concomitant elevations in NO. This might prove more efficacious than simply inhibiting the enzyme using classical inhibitors. Importantly, a recent study (EXACT-HF) has shown a trend for reduced HF re-hospitalisations in those with XOR inhibition via allopurinol; it has been suggested that greater benefits might be seen if these effects are coupled with NO delivery.

Research Hypothesis and Aims: We aim to investigate whether dietary inorganic nitrate provides benefit in patients with HF. We will determine whether inorganic nitrate delivery by elevating nitrite, delivers substrate to XOR resulting in a two-fold benefit: increasing NO production, whilst concomitantly reducing superoxide and uric acid levels.

Plan of Investigation: a randomised double-blind placebo-controlled parallel two-limb study in New York Heart Association (NHYA) class II-III HF patients. Patients with left ventricular ejection fraction (LVEF) <50% and elevated NT-proBNP/ BNP levels will be enrolled and stratified by degree of hyperuricaemia. 92-patients will receive a once daily dose of nitrate-rich beetroot juice (versus nitrate-deplete beetroot juice) for 12-weeks. The study is powered for significant reductions in hyperuricaemia. Powered secondary outcomes include circulating nitrite/nitrate levels, nitrite reductase activity, and a difference in LVEF from baseline by contrast echocardiography. A number of mechanistic exploratory outcomes will also be reported, including assessments of oxidative stress, erythrocytic XOR activity, 6-minute walk test, quality of life questionnaire and levels of NT-proBNP/BNP as surrogate measures of cardiac dysfunction.

Benefits: This trial if positive will identify a new, safe and easy-to-deliver therapeutic option for HF patients. The NHS would benefit by providing a new inexpensive pharmacotherapy for a disease with significant unmet need and increasing burden to the health service.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosed with heart failure with reduced ejection fraction on the basis of:

   1. LVEF ≤50% as assessed by Echocardiography (or cardiac MRI)
   2. raised BNP and/or NT-proBNP levels placing patients in the "high risk" category, to ensure heart failure is the cause of symptoms:

      * stable heart failure: NT-proBNP >600pg/mL and BNP >150pg/mL
      * hospitalisation within 12 months: NT-proBNP >400pg/mL and BNP >100pg/mL
3. NYHA Class II-III symptoms
4. On optimally-tolerated, stable (>12 weeks) prognostic medical therapy (beta-blocker, ACE-inhibitor or ARB, mineralocorticoid therapy if deemed necessary)
5. No heart failure-related hospitalisation for >12 weeks
6. Clinic systolic blood pressure ≥95mmHg
7. Able and willing to give written informed consent

The intervention with dietary nitrate is intentionally designed to be in addition to the patient's own lifestyle. There will be no restrictions placed on diet, anti-oxidant supplements or prescription medications, other than those listed in the exclusion criteria below.

Exclusion Criteria:

1. Use of anti-bacterial mouthwash or tongue scrapes (current or unwillingness to cease such mouthcare for at least one month prior to entering the study, and for the duration of the trial) as this interrupts the enterosalivary circuit and thus prevents the bioactivity of nitrate
2. History of recurrent symptomatic gout or current treatment with xanthine oxidase inhibitors for hyperuricaemia
3. Concomitant use of long acting organic nitrates or phosphodiesterase inhibitors (not including on an as required basis)
4. Angina at CCS Class III/IV, requiring regular use of sublingual GTN (considered >twice/week), or awaiting revascularisation
5. If LVEF in the range 40-50%, impaires systolic function secondary to uncorrected valve disease, primary pulmonary hypertension, active myocarditis, constrictive pericarditis, restrictive cardiomyopathy or hypertrophic cardiomyopathy
6. Renal failure with eGFR<30 at screening
7. History of symptomatic renal stone disease
8. Current life-threatening condition that might prevent a patient-subject completing the study
9. Allergy to SonoVue Echo contrast
10. Pregnancy, breast feeding or planned pregnancy
11. Anaemia, defined as Haemaglobin <80g/L
12. Subjects with any acute infection, or recent systemic antibiotics (oral or intravenous) within 3 months of screening, or significant trauma (burns, fractures)
13. The subject has a three-month prior history of regular alcohol consumption exceeding an average weekly intake of > 28 units (or an average daily intake of greater than 3 units) for males, or an average weekly intake of > 21 units (or an average daily intake of greater than 2 units) for females. 1 unit is equivalent to a half-pint (284mL) of beer/lager; 25mL measure of spirits or 125mL of wine
14. Mobility thought to be restricted significantly by other illnesses apart from heart failure
15. Any other subject whom the Investigator deems unsuitable for the study (e.g. due to other medical reasons, laboratory abnormalities, expected study medication noncompliance, or subject's unwillingness to comply with all study-related study procedures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2025-01-07 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Change in serum uric acid levels | 12 +/- 2 weeks
  Uric acid is a prognostic marker in patients with heart failure. The intervention proposed acts on the enzyme, xanthine oxidoreductase (XOR), that produces uric acid. We will therefore measure the change in serum uric acid level from baseline to assess whether dietary nitrate treatment decreases hyperuricaemia. We will stratify uric acid levels and undertake analysis between strata.

SECONDARY OUTCOMES:
Changes in plasma nitrate | 12 +/- 2 weeks
  We will measure the change in nitrate levels in plasma using ozone chemiluminescence, which measures the consumed dose of inorganic nitrate consumed, as the first step in the enterosalivary circuit.
Changes in plasma nitrite | 12 +/- 2 weeks
  We will measure the change in nitrite levels in plasma using ozone chemiluminescence, measuring the conversion of nitrate to nitrite which the enzyme XOR uses to form the biologically active metabolite, nitric oxide.
Changes in cGMP as a marker for Nitric Oxide | 12 +/- 2 weeks
  We will measure the change in cGMP levels using an ELISA assay, as a stable and measurable surrogate of the biologically active product, nitric oxide.
Changes in cardiac pump function | 12 +/- 2 weeks
  Using contrast Echocardiography, we will measure the change in left ventricular ejection fraction from baseline following intervention.

OTHER OUTCOMES:
Changes in markers of oxidative stress: MDA | 12 +/- 2 weeks
  Measured using ELISA and used collectively with oxidised LDL and TBAR assays to determine oxidative stress
Changes in markers of oxidative stress: oxidised LDL | 12 +/- 2 weeks
  Measured using ELISA and used collectively with MDA and TBAR assays to determine oxidative stress
Changes in markers of oxidative stress: TBAR | 12 +/- 2 weeks
  Measured using ELISA and used collectively with oxidised LDL and MDA assays to determine oxidative stress
Measure of red blood cell XOR activity | 12 +/- 2 weeks
  We will measure expression and activity of XOR by red blood cells, as a marker of both nitrite reductase capacity as well as hyperuricaemia.
Changes in blood pressure | 12 +/- 2 weeks
  Analysis of 24-hour blood pressure monitoring
Change in NT-proBNP | 12 +/- 2 weeks
  Analysis of this important natriuretic peptide
Change in BNP | 12 +/- 2 weeks
  Analysis of this important natriuretic peptide
Change in high sensitivity C-Reactive Protein | 12 +/- 2 weeks
  Analysis of the highly sensitive marker of inflammation
Change in lipid levels (LDL, triglycerides, HDL, total cholesterol) | 12 +/- 2 weeks
  Analysis of lipids
Contrast Echocardiography: ventricular function | 12 +/- 2 weeks
  Measurement of cardiac ventricular function using cardiac MRI (ejection fraction)
Contrast Echocardiography: ventricular volumes | 12 +/- 2 weeks
  Measurement of cardiac ventricular volumes using cardiac MRI
Contrast Echocardiography: wall stress | 12 +/- 2 weeks
  Assessment of left ventricular wall stress
Changes in resting cardiac electrical activity | 12 +/- 2 weeks
  As determined by electrocardiogram analysis
6-minute Walk Test | 12 +/- 2 weeks
  Functional assessment of exercise capacity
Minnesota Living with Heart Failure Quality of Life Questionnaire | 12 +/- 2 weeks
  Qualitative analysis of quality of life
Stratification by Type II Diabetes Mellitus | 12 +/- 2 weeks
  All results will be stratified by the pre-existing diagnosis of Type II Diabetes Mellitus to determine whether this additional cause of oxidative stress impacts on the ability of inorganic nitrate to recover function in patients with heart failure
Evidence of active dental caries | 12 +/- 2 weeks
  Pre-specified sub-group analyses by dental disease
Measurement of methaemaglobinaemia | 12 +/- 2 weeks
  Safety measure

CONTACTS AND LOCATIONS:
Overall Officials: Dr Simon Woldman, MD FRCP FESC, Principal Investigator — Fellow of the Royal College of Physicians and Fellow of the European Society of Cardiology; Dr Ceri Davies, MD FRCP FESC, Principal Investigator — Fellow of the Royal College of Physicians and Fellow of the European Society of Cardiology; Prof Amrita Ahluwalia, BSc PhD, Study Chair — William Harvey Research Institute, Queen Mary University of London
Locations (1):
- Queen Mary University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not applicable - no plans to share IPD

REFERENCES:
- [Background] Kapil V, Khambata RS, Robertson A, Caulfield MJ, Ahluwalia A. Dietary nitrate provides sustained blood pressure lowering in hypertensive patients: a randomized, phase 2, double-blind, placebo-controlled study. Hypertension. 2015 Feb;65(2):320-7. doi: 10.1161/HYPERTENSIONAHA.114.04675. Epub 2014 Nov 24. PMID 25421976
- [Background] Velmurugan S, Gan JM, Rathod KS, Khambata RS, Ghosh SM, Hartley A, Van Eijl S, Sagi-Kiss V, Chowdhury TA, Curtis M, Kuhnle GG, Wade WG, Ahluwalia A. Dietary nitrate improves vascular function in patients with hypercholesterolemia: a randomized, double-blind, placebo-controlled study. Am J Clin Nutr. 2016 Jan;103(1):25-38. doi: 10.3945/ajcn.115.116244. Epub 2015 Nov 25. PMID 26607938
- [Background] Jones DA, Pellaton C, Velmurugan S, Rathod KS, Andiapen M, Antoniou S, van Eijl S, Webb AJ, Westwood MA, Parmar MK, Mathur A, Ahluwalia A. Randomized phase 2 trial of intracoronary nitrite during acute myocardial infarction. Circ Res. 2015 Jan 30;116(3):437-47. doi: 10.1161/CIRCRESAHA.116.305082. Epub 2014 Dec 15. PMID 25512434
- [Background] Givertz MM, Anstrom KJ, Redfield MM, Deswal A, Haddad H, Butler J, Tang WH, Dunlap ME, LeWinter MM, Mann DL, Felker GM, O'Connor CM, Goldsmith SR, Ofili EO, Saltzberg MT, Margulies KB, Cappola TP, Konstam MA, Semigran MJ, McNulty SE, Lee KL, Shah MR, Hernandez AF; NHLBI Heart Failure Clinical Research Network. Effects of Xanthine Oxidase Inhibition in Hyperuricemic Heart Failure Patients: The Xanthine Oxidase Inhibition for Hyperuricemic Heart Failure Patients (EXACT-HF) Study. Circulation. 2015 May 19;131(20):1763-71. doi: 10.1161/CIRCULATIONAHA.114.014536. Epub 2015 Apr 14. PMID 25986447
- [Background] Khambata RS, Ghosh SM, Rathod KS, Thevathasan T, Filomena F, Xiao Q, Ahluwalia A. Antiinflammatory actions of inorganic nitrate stabilize the atherosclerotic plaque. Proc Natl Acad Sci U S A. 2017 Jan 24;114(4):E550-E559. doi: 10.1073/pnas.1613063114. Epub 2017 Jan 5. PMID 28057862